CLINICAL TRIAL: NCT02227550
Title: An Investigator-driven, Prospective, Parallel-group, Randomised, Open, Blinded Outcome Assessment (PROBE), Multi-centre Trial to Determine the Optimal Anticoagulation Therapy for Patients Untergoing Catheter Ablation of Atrial Fibrillation
Brief Title: Apixaban During Atrial Fibrillation Catheter Ablation: Comparison to Vitamin K Antagonist Therapy
Acronym: AXAFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFNET 5 AXAFA; 2014-002442-45 (EudraCT Number)
Record Dates: First submitted 2014-06-27; First posted 2014-08-28 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrilal fibrillation; anticoagulation; prevention of peri-procedural complication; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — acarboxyprothrombin; Warfarin; Phenprocoumon; fluindione; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental): Xa group: factor Xa inhibitor Apixaban min. 30 days 5 mg twice daily (fix dose)
  Interventions: Drug: Apixaban
- Vitamin K antagonist (Active Comparator): VKA group: any Vitamin K antagonist (VKA), INR 2-3 , min. 30 days prescribed as in clinical routine
  Interventions: Drug: Vitamin K antagonist

INTERVENTIONS:
Drug: Vitamin K antagonist — any locally used VKA, INR 2-3, min. 30 days according to aplicable medical guidelines and local clinical routin
  Other Names: warfarin; phenprocoumon; acecoumaril; fluindione
  Arms: Vitamin K antagonist
Drug: Apixaban — factor Xa inhibitor Apixaban min. 30 days 5 mg twice daily (fix dose) dose reduction Apixaban 2,5 mg twice daily in patients who fulfill tow of the following criteria at the time of randomisation: chronic kidney disease (serum creatine >= 1.5 mg/dl (133mM), <= 60 kg body weight or age >= 80 years.
  Other Names: BMS-562247
  Arms: Apixaban

SUMMARY:
Study objective is to demonstrate that anticoagulation with the direct factor Xa inhibitor apixaban is not less safe than Vitamin-K-antagonists (VKA) therapy in patients undergoing catheter ablation of non-valvular AF in the prevention of peri-procedural complications.

The AXAFA trial will compare peri-ablational treatment with apixaban to peri-ablational treatment wit VKA in a randomized trial of patients undergoing catheter ablation of atrial fibrillation (AF).

DETAILED DESCRIPTION:
AXAFA is an open-label trial designed to evaluate the safety and efficacy of two types of anticoagulant therapy, VKA therapy and therapy with the direct factor Xa inhibitor apixaban, in patients undergoing scheduled catheter ablation for AF. All patients will undergo the ablation procedure after pre-treatment with an anticoagulant (either apixaban in the "Xa group" or a vitamin K antagonist in the "VKA group").

Patients can undergo catheter ablation within the trial after at least 30 days of continuous effective anticoagulation. Ablation can be performed earlier when or timely after exclusion of atrial thrombi have been excluded by a clinically indicated by transthoracic echocardioggram (TEE). After TEE continuous effective anticoagulation must be ensured until the end of the trial.

In the MRI-substudy will be explored wether novel oral anticoagulants (NOAC) have the potential to reduce clinically silent brain lesions after catheter ablation of AF.

ELIGIBILITY:
Inclusion Criteria:

I1. Non-valvular AF (ECG-documented) with a clinical indication for catheter ablation

I2. Clinical indication to undergo catheter ablation on continuous anticoagulant therapy

I3. Presence of at least one of the CHADS2 stroke risk factors

* Stroke or TIA
* age ≥ 75 years,
* hypertension, defined as chronic treatment for hypertension, estimated need for continuous antihypertensive therapy or resting blood pressure > 145/90 mm Hg,
* diabetes mellitus,
* symptomatic heart failure (NYHA ≥ II).

I4. Age ≥ 18 years

I5. Provision of signed informed consent

Exclusion Criteria:

General exclusion criteria

E1. Any disease that limits life expectancy to less than 1 year

E2. Participation in another clinical trial, either within the past two months or still ongoing

E3. Previous participation in AXAFA

E4. Pregnant women or women of childbearing potential not on adequate birth control: only women with a highly effective method of contraception (oral contraception or intra-uterine device) or sterile women can be randomised.

E5. Breastfeeding women

E6. Drug abuse or clinically manifest alcohol abuse

E7. Any stroke within 14 days before randomisation

E8. Coadministration with drugs that are strong dual inhibitors of cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp) or strong dual inducers of CYP3A4 and P-gp (Appendix VIII).

Exclusion criteria related to a cardiac condition

E9. Valvular AF (as defined by the focussed update of the ESC guidelines on AF, i.e. severe mitral valve stenosis, mechanical heart valve). Furthermore, patients who underwent mitral valve repair are not eligible for AXAFA.

E10. Any previous ablation or surgical therapy for AF

E11. Cardiac ablation therapy for any indication (catheter-based or surgical) within 3 months prior to randomisation

E12. Clinical need for "triple therapy" (combination therapy of clopidogrel, acetylsalicylic acid, and oral anticoagulation)

E13. Other contraindications for use of VKA or apixaban

E14. Documented atrial thrombi less than 3 months prior to randomisation.

Exclusion criteria based on laboratory abnormalities

E15. Severe chronic kidney disease with an estimated glomerular filtration rate (GFR) < 15 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2014-12; Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
death and serious cardiovascular events | appr. 4 months
  A composite of all-cause death, stroke (ischemic stroke, subarachnoid haemorrhage and haemorrhagic stroke), and major bleeding events, def.as BARC 2 or higher

SECONDARY OUTCOMES:
any bleeding event | appr. 4 months
  number
major bleeding events acc. to the ISTH and TIMI definitions | appr. 4 months
  number
strokes, other systemic embolic events and all-cause death | appr. 4 month
  number
time from randomisation to ablation | appr. 4 months
  number of days
nights spent in hospital after ablation | appr. 4 months
  number
health-care related cost calculation | appr. 4 months
hospitalizations for cardiovascular reasons | appr. 4 months
  number
Treatment duration prior to ablation and total time on oral anticoagulation | appr. 4 months
  number of days
patients with clinically indicated TEE | appr. 4 months
  number of patients
ACT during ablation | during ablation
  Active clotting measurements
recurrent Atrial Fibrillation (AF) | appr. 4 months
  time to recurrent AF
rhythm status at the end of follow-up | end of follow-up
  rythm status documented by 24 hour Holter ECG
vascular access complications leading to prolongation of in-hospital stay or specific therapy | appr. 4 months
  number of events
Quality-of-life changes | baseline to 3 month follow-up
  questionaire
cognitive function change | baseline to 3 month follow-up
  questionaire
clinically "silent" MRI-detected brain lesions | within 48 hours after ablation procedures
  prevalence (MRI-substudy)
Impact of ablation-associated clinically overt strokes or MRI-detected bus clincally "silent" acute brain lesions on cognitive function after ablation | appr. 4 months
  MRI-substudy

CONTACTS AND LOCATIONS:
Overall Officials: Paulus Kirchhof, Professor, Principal Investigator — University of Birmingham Centre for Cardiovascular Scienes, UK and University Hospital Muenster, Germany
Locations (13):
- United States (5):
  - Montefiore Medical Center, New York, New York
  - Hospital of the University of Pennsyvlania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Sentara Cariovascular Research Insititute, Norfolk, Virginia
- 4 Sites, Different, Austria
- 5 Sites, Different, Belgium
- 5 Sites, Different, Denmark
- 13 Sites, Different, Germany
- 4 Sites, Different, Italy
- 6 Sites, Different, Netherlands
- 3 Sites, Different, Spain
- 4 Sites, Different, United Kingdom

REFERENCES:
- [Background] Di Biase L, Callans D, Haeusler KG, Hindricks G, Al-Khalidi H, Mont L, Cosedis Nielsen J, Piccini JP, Schotten U, Kirchhof P. Rationale and design of AXAFA-AFNET 5: an investigator-initiated, randomized, open, blinded outcome assessment, multi-centre trial to comparing continuous apixaban to vitamin K antagonists in patients undergoing atrial fibrillation catheter ablation. Europace. 2017 Jan;19(1):132-138. doi: 10.1093/europace/euw368. PMID 28130378
- [Derived] Haeusler KG, Eichner FA, Heuschmann PU, Fiebach JB, Engelhorn T, Callans D, De Potter T, Debruyne P, Scherr D, Hindricks G, Al-Khalidi HR, Mont L, Kim WY, Piccini JP, Schotten U, Themistoclakis S, Di Biase L, Kirchhof P. Detection of brain lesions after catheter ablation depends on imaging criteria: insights from AXAFA-AFNET 5 trial. Europace. 2023 Dec 6;25(12):euad323. doi: 10.1093/europace/euad323. PMID 37897713
- [Derived] Haeusler KG, Eichner FA, Heuschmann PU, Fiebach JB, Engelhorn T, Blank B, Callans D, Elvan A, Grimaldi M, Hansen J, Hindricks G, Al-Khalidi HR, Mont L, Nielsen JC, Piccini JP, Schotten U, Themistoclakis S, Vijgen J, Di Biase L, Kirchhof P. MRI-Detected Brain Lesions and Cognitive Function in Patients With Atrial Fibrillation Undergoing Left Atrial Catheter Ablation in the Randomized AXAFA-AFNET 5 Trial. Circulation. 2022 Mar 22;145(12):906-915. doi: 10.1161/CIRCULATIONAHA.121.056320. Epub 2022 Feb 9. PMID 35135308
- [Derived] Zink MD, Chua W, Zeemering S, di Biase L, Antoni BL, David C, Hindricks G, Haeusler KG, Al-Khalidi HR, Piccini JP, Mont L, Nielsen JC, Escobar LA, de Bono J, Van Gelder IC, de Potter T, Scherr D, Themistoclakis S, Todd D, Kirchhof P, Schotten U. Predictors of recurrence of atrial fibrillation within the first 3 months after ablation. Europace. 2020 Sep 1;22(9):1337-1344. doi: 10.1093/europace/euaa132. PMID 32725107